CLINICAL TRIAL: NCT03896399
Title: Laparoscopic Ischemic Conditioning Prior to Esophagectomy in Patients With Esophageal Cancer and Arterial Calcifications
Brief Title: Laparoscopic Ischemic Conditioning Prior to Esophagectomy
Acronym: ISCON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Richard van Hillegersberg, Professor, surgeon, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL67819.041.18
Record Dates: First submitted 2019-03-20; First posted 2019-04-01 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Esophagectomy; Ischemic conditioning
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic ischemic conditioning followed by esophagectomy (Experimental): All included patients will receive a laparoscopic ischemic conditioning followed by an esophagectomy after an interval of 12-18 days.
  Interventions: Procedure: Laparoscopic ischemic conditioning followed by esophagectomy

INTERVENTIONS:
Procedure: Laparoscopic ischemic conditioning followed by esophagectomy — All included patients will receive a laparoscopic ischemic conditioning followed by an esophagectomy after an interval of 12-18 days.

SUMMARY:
This is a two center phase II prospective single-arm safety and feasibility trial for 20 patients with resectable esophageal carcinoma with an increased risk for anastomotic leakage, as based upon UCS and NASCET calcification scores on pre-op CT-scan. In these patients, laparoscopic ischemic conditioning is performed 12-18 days before an Ivor-Lewis esophagectomy. The primary outcome is all complications grade 2 and higher (Clavien-Dindo classification) occurring during or after the laparoscopic ischemic conditioning. Secondary outcomes are complications after the esophagectomy, and the induction of angiogenesis by biomarkers of microcirculation and redistribution of blood flow by measurement of indocyanine green (ICG) fluorescence angiography.

DETAILED DESCRIPTION:
Rationale:

Anastomotic leakage is the most important surgical complication following esophagectomy for esophageal cancer, leading to increased morbidity and mortality. A major cause of leakage is impaired healing due to ischemia of the gastric tube that is used for reconstruction of the gastrointestinal tract. Calcifications of the aorta or stenosis of the celiac trunk on pre-operative CT scan have been shown to be associated with an increased risk of anastomotic leakage. So far, no individualized treatment has been initiated for this selected group of patients. Laparoscopic ischemic conditioning (ISCON) of the gastric tube aims to increase perfusion at the anastomotic site by redistribution of the gastric blood flow and/or induction of angiogenesis. This is achieved by occlusion of the supplying gastric arteries except for the right gastroepiploic artery during a separate intervention prior to esophagectomy. Of note, these arteries would also be occluded during conventional esophagectomy, but with laparoscopic ISCON they are occluded at an earlier moment in time during a separate intervention. Retrospective studies have demonstrated the safety of this technique. Prospective studies have not yet been performed.

Primary objective:

Assess the safety and feasibility of laparoscopic ISCON 12-18 days prior to esophagectomy for esophageal cancer in patients with arterial calcifications.

Study design:

Two center phase II prospective single-arm safety and feasibility trial.

Study population:

Patients with resectable esophageal carcinoma (cT1-4a, N0-3, M0) with "major calcifications" of the thoracic aorta (UCS) and any additional calcification or stenosis of the celiac axis (modified NASCET score) on preoperative CT scan, who are planned to undergo esophagectomy.

Intervention:

Laparoscopic ISCON followed by esophagectomy after an interval of 12-18 days.

Primary outcome:

all complications grade 2 and higher (Clavien-Dindo classification) occurring during or after operation 1 (laparoscopic ISCON) and before operation 2 (esophagectomy).

Secondary outcomes:

secondary outcomes with regard to operation 1 (laparoscopic ISCON) are the duration of the procedure, blood loss, day of discharge postoperatively and grade 1 complications. Secondary outcomes with regard to operation 2 (esophagectomy) are anastomotic leakage rate, all other grade 3b or higher complications and 30 day mortality. Further secondary endpoints are the induction of angiogenesis by biomarkers of microcirculation and redistribution of blood flow by measurement of indocyanine green (ICG) fluorescence angiography.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

the additional burden for the patient consists of an extra operation of approximately 40 minutes during which laparoscopic ISCON will be performed, prior to the planned esophagectomy. We would classify the current study as medium risk. Potential benefits in comparison to current standard treatment are a reduced risk of anastomotic leakage and severity of anastomotic leakage. Potential risks are complications following operation 1 (laparoscopic ISCON). Mainly, based upon prior experience, we expect gastroparesis to occur in 25% of patients. Patients with gastroparesis have an increased risk of aspiration and will require a stomach emptying by nasogastric tube and nasojejunal tube feeding till the performance of operating 2 (esophagectomy).

ELIGIBILITY:
Inclusion criteria:

* Histologically proven adenocarcinoma (AC) or squamous cell carcinoma (SCC) of the esophagus or gastroesophageal junction (GEJ)
* Planned to undergo transthoracic esophagectomy or transhiatal esophagectomy
* Preoperative computed tomography (CT)
* Vascular arterial changes: "major calcifications" of the thoracic aorta according to the "Uniform calcification score" (UCS) and or a stenosis of the celiac axis according to the "modified NASCET score". (Appendix 1 and 2) (7,17)
* ASA I-III
* European Clinical Oncology Group (ECOG) performance status of 0,1 or 2
* Age > 17
* Written informed consent

Exclusion criteria:

* Not able to undergo study treatment.
* Metastatic disease (M1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a grade 2 or higher complication after laparoscopic ischemic conditioning | Occuring after operation 1(laparosocpic ISCON), but before operation 2 (esophagectomy). This time-frame is usually 13-15 days.
  Complications grade 2 and higher (Clavien-Dindo classification)

SECONDARY OUTCOMES:
Number of participants with a grade 1 complication after operation 1 (laparoscopic ISCON) | Occuring after operation 1(laparosocpic ISCON), but before operation 2 (esophagectomy). This time-frame is usually 13-15 days.
  Grade 1 complications after operation 1 (laparoscopic ISCON)
Duration of operation 1 (laparoscopic ISCON) | During operation 1
  Duration of operation 1 (laparoscopic ISCON)
Bloodloss during operation 1 (laparoscopic ISCON) | During operation 1
  Bloodloss during operation 1 (laparoscopic ISCON)
Day of discharge after operation 1 (laparoscopic ISCON) | After operation 1, usually on the third post-operative day
  Day of discharge after operation 1 (laparoscopic ISCON)
Number of participants with anastomotic leakage after operation 2 (esophagectomy) | Within 30 days after operation 2
  Anastomotic leakage after operation 2 (esophagectomy)
Number of participants with grade 3b or higher complications after operation 2 (esophagectomy) | Within 30 days after operation 2
  Grade 3b (Clavien-Dindo classification) or higher complications after operation 2 (esophagectomy)
Number of participants with 30 day mortality after operation 2 (esophagectomy) | Within 30 days after operation 2
  30 day mortality after operation 2 (esophagectomy)
Induction of angiogenesis in tissue | Biopsies are taken at the start, or within 24 hours of operation 1 and operation 2. In addition, the anastomoc donut or tip of gastric tube is collected during operation 2 (esophagectomy) after formation of the anastomosis.
  Paraffin embedded sections (10µm) will be stained by immunohistochemistry against CD31 (vessel density) or smooth-muscle-actin positive pericytes to characterize vascularity
Induction of angiogenesis by biomarkers of microcirculation | Peripheral blood is taken at the start, or within 24 hours of operation 1
  A cytokine profile will be measured in the peripheral blood, consisting of VEGF, IL-8, IL-6, TNF-alpha and Ang-2
Redistribution of blood flow by measurement of indocyanine green (ICG) fluorescence angiography | During operation 1 and during operation 2 (esophagectomy)
  Redistribution of blood flow by measurement of indocyanine green (ICG)

CONTACTS AND LOCATIONS:
Overall Officials: Richard van Hillegersberg, MD, PhD, Principal Investigator — University Medical Center Utrecht, dept. of Surgery; Wolfgang Schröder, MD, PhD, Principal Investigator — University Hospital of Cologne, department of Surgery
Locations (2):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
This will be published
Supporting Information: Study Protocol, SAP
Time Frame: The protocol will be published in an international journal after the start of the study
Access Criteria: The protocol will be accessibel from the journal in which it will be published

REFERENCES:
- [Derived] Veen AV, Schiffmann LM, de Groot EM, Bartella I, de Jong PA, Borggreve AS, Brosens LAA, Santos DPD, Fuchs H, Ruurda JP, Bruns CJ, van Hillegersberg R, Schroder W. The ISCON-trial protocol: laparoscopic ischemic conditioning prior to esophagectomy in patients with esophageal cancer and arterial calcifications. BMC Cancer. 2022 Feb 5;22(1):144. doi: 10.1186/s12885-022-09231-x. PMID 35123419